CLINICAL TRIAL: NCT05498428
Title: A Phase 2, Open-Label, Parallel Cohort Study of Subcutaneous Amivantamab in Multiple Regimens in Patients With Advanced or Metastatic Solid Tumors Including EGFR-mutated Non-Small Cell Lung Cancer
Brief Title: A Study of Amivantamab in Participants With Advanced or Metastatic Solid Tumors Including Epidermal Growth Factor Receptor (EGFR)-Mutated Non-Small Cell Lung Cancer
Acronym: PALOMA-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109264; 61186372NSC2002 (Other: Janssen Research & Development, LLC); 2022-000526-21 (EudraCT Number); 2023-505065-91-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; lazertinib; Carboplatin; Pemetrexed; N(4)-oleylcytosine arabinoside; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1(Exon19del/Exon21 L858R NSCLC, 1L, Previously Untreated): Amivantamab (Q2W) + Lazertinib (Experimental): Participants with treatment-naive locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring an epidermal growth factor receptor (EGFR) exon 19 deletion (exon19del) or exon 21 leucine 858 to arginine substitution (exon 21 L858R) mutation, will receive amivantamab SC-CF injection, 1600 milligrams (mg) or 2240 mg if body weight is greater than or equal to (>=) 80 kilograms (kg), on Cycle 1 Days 1, 8, 15, and 22 and on Days 1 and 15 of each subsequent 28-day cycle, starting with Cycle 2, along with lazertinib 240 mg orally once daily. Eligible participants will be given an option to enter long-term extension (LTE) phase and may continue to receive access to study treatment(s) within the study by transferring to the Drug Access (DA)-LTE Phase.
  Interventions: Drug: Amivantamab; Drug: Lazertinib
- Cohort 2(Exon20 NSCLC,1L, Previously Untreated): Amivantamab (Q3W) + Chemotherapy (Experimental): Participants with treatment-naive locally advanced or metastatic NSCLC harboring an EGFR exon20ins mutation will receive Amivantamab SC-CF injection 1600 mg or 2240 mg if body weight is >=80 kg on Cycle 1 Day 1, 2400 mg or 3360 mg if body weight is >=80 kg on Cycle 1 Day 8 and 15 and on Day 1 of each subsequent 21-day cycle, starting with Cycle 2 along with pemetrexed 500 milligrams per meter square (mg/m^2) as intravenous (IV) infusion (with vitamin supplementation) on Day 1 of each 21-day cycle and IV infusion carboplatin area under the concentration-time curve 5 milligrams per milliliters (mg/mL) per minute (AUC 5) maximum 750 mg on Day 1 of each 21-day cycle, for up to 4 cycles. Eligible participants will be given an option to enter LTE phase and may continue to receive access to study treatment(s) within the study by transferring to the DA-LTE Phase.
  Interventions: Drug: Amivantamab; Drug: Carboplatin; Drug: Pemetrexed
- Cohort 3(Exon19del/Exon21 L858R NSCLC,2L,Post Osimertinib):Amivantamab(Q3W)+Lazertinib+Chemotherapy (Experimental): Participants with locally advanced or metastatic NSCLC harboring an EGFR exon19del or exon 21 L858R mutation who have experienced disease progression on or after treatment with a third-generation EGFR TKI (osimertinib), will receive amivantamab SC-CF injection 1600 mg or 2240 mg if body weight is >=80 kg on Cycle 1 Day 1, 2400 mg or 3360 mg if body weight is >=80 kg on Cycle 1 Day 8 and 15 and on Day 1 of each subsequent 21-day cycle starting with Cycle 2; in combination with IV infusion carboplatin area under the concentration-time curve 5 mg/mL per minute (AUC 5) maximum 750 mg on Day 1 of each 21-day cycle, for up to 4 cycles; and pemetrexed 500 mg/m^2 as an IV infusion (with vitamin supplementation) on Day 1 of each 21-day until disease progression. Lazertinib 240 mg orally once daily starting Cycle 5 Day 1 when carboplatin is complete or sooner if carboplatin discontinued earlier than Cycle 4. Eligible participants will be given an option to enter LTE phase and DA-LTE Phase.
  Interventions: Drug: Amivantamab; Drug: Lazertinib; Drug: Carboplatin; Drug: Pemetrexed
- Cohort 3b(Exon19del/Exon21 L858R NSCLC, 2L, Post Osimertinib): Amivantamab (Q3W)+Chemotherapy (Experimental): Participants with locally advanced or metastatic NSCLC harboring an EGFR exon19del or exon 21 L858R mutation who have experienced disease progression on or after treatment with a third-generation EGFR TKI (osimertinib), will receive amivantamab SC-CF injection 1600 mg or 2240 mg if body weight is >=80 kg on Cycle 1 Day 1, 2400 mg or 3360 mg if body weight is >=80 kg on Cycle 1 Day 8 and 15 and on Day 1 of each subsequent 21-day cycle starting with Cycle 2; in combination with IV infusion carboplatin area under the concentration-time curve 5 mg/mL per minute (AUC 5) maximum 750 mg on Day 1 of each 21-day cycle, for up to 4 cycles; and pemetrexed 500 mg/m^2 as an IV infusion (with vitamin supplementation) on Day 1 of each 21-day until disease progression. Eligible participants will be given an option to enter LTE phase and may continue to receive access to study treatment(s) within the study by transferring to the DA-LTE Phase.
  Interventions: Drug: Amivantamab; Drug: Carboplatin; Drug: Pemetrexed
- Cohort 4(Previously Treated with Amivantamab IV): Switch from Amivantamab IV to SC-CF (Q2W) (Experimental): Participants who were previously on amivantamab IV once every 2 weeks (Q2W) regimen as part of standard of care, for at least 8 weeks, either as monotherapy or combination with lazertinib, will receive amivantamab SC-CF injection 1600 mg and 2240 mg if body weight is greater than or equal to 80 kg. Participants who continue to benefit from study treatments, as determined by their investigator, may shift to the drug access (DA)-LTE phase.
  Interventions: Drug: Amivantamab; Drug: Lazertinib
- Cohort 5(Exon19del/Exon21 L858R NSCLC, 1L, Previously Untreated): Amivantamab (Q4W) + Lazertinib (Experimental): Participants with treatment-naïve locally advanced or metastatic NSCLC harboring an EGFR Exon19del or Exon 21 L858R mutation will receive amivantamab SC-CF induction with 1,600 mg (or 2,240 mg if BW >=80 kg) on Cycle 1 Days 1, 8, 15, and 22, starting with Cycle 2 on Day 1 of each next 28-day cycle, amivantamab SC-CF (160 mg/mL co-formulated with rHuPH20) by manual injection at 3,520 mg (or 4,640 mg if BW >=80 kg); along with lazertinib 240 mg by mouth once daily from Cycle 1 Day 1. Eligible participants will be given an option to enter LTE phase and may continue to receive access to study treatment(s) within the study by transferring to the DA-LTE Phase.
  Interventions: Drug: Amivantamab; Drug: Lazertinib
- Cohort6(Exon19del/Exon21L858R,NSCLC1L,PreviouslyUntreated):Amivantamab(Q2W)+Lazertinib+Anticoagulant (Experimental): Participants with treatment-naive locally advanced or metastatic NSCLC harboring an EGFR Exon19del or Exon 21 L858R mutation treated will receive will receive amivantamab SC-CF injection, 1600 milligrams (mg) and 2240 mg if body weight is greater than or equal to (>=) 80 kilograms (kg), on Cycle 1 Days 1, 8, 15, and 22 and on Days 1 and 15 of each subsequent 28-day cycle, starting with Cycle 2, along with lazertinib 240 mg orally once daily from Cycle 1 Day 1. Participants will additionally take prophylactic anticoagulation with a direct oral anticoagulant (DOAC) or a low molecular weight heparin (LMWH) for the first four months of study treatment (from Day 1 through Day 120) with the combination of amivantamab and lazertinib. Eligible participants will be given an option to enter LTE phase and may continue to receive access to study treatment(s) within the study by transferring to the DA-LTE Phase.
  Interventions: Drug: Amivantamab; Drug: Lazertinib; Drug: Direct Oral Anticoagulant (DOAC); Drug: Low Molecular Weight Heparin (LMWH)
- Cohort 7(Exon19del/Exon21 L858R NSCLC,2L,Post Amivantamab+Lazertinib):Amivantamab(Q3W)+Chemotherapy (Experimental): Participants with locally advanced or metastatic NSCLC harboring an EGFR exon19del or exon 21 L858R mutation who have experienced disease progression on or after the combination of amivantamab and lazertinib will receive amivantamab SC-CF injection 1600 mg or 2240 mg if body weight is >=80 kg on Cycle 1 Day 1, 2400 mg or 3360 mg if body weight is >=80 kg on Cycle 1 Day 8 and 15 and on Day 1 of each subsequent 21-day cycle starting with Cycle 2; in combination with IV infusion carboplatin area under the concentration-time curve 5 mg/mL per minute (AUC 5) maximum 750 mg on Day 1 of each 21-day cycle, for up to 4 cycles; and pemetrexed 500 mg/m^2 as an IV infusion (with vitamin supplementation) on Day 1 of each 21-day until disease progression. Eligible participants will be given an option to enter LTE phase and may continue to receive access to study treatment(s) within the study by transferring to the DA-LTE Phase.
  Interventions: Drug: Amivantamab; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Amivantamab — Amivantamab will be administered subcutaneously by manual injection.
  Other Names: JNJ-61186372
Drug: Lazertinib — Lazertinib will be administered as an oral tablet.
  Other Names: JNJ-73841937; YH25448
  Arms: Cohort 1(Exon19del/Exon21 L858R NSCLC, 1L, Previously Untreated): Amivantamab (Q2W) + Lazertinib; Cohort 3(Exon19del/Exon21 L858R NSCLC,2L,Post Osimertinib):Amivantamab(Q3W)+Lazertinib+Chemotherapy; Cohort 4(Previously Treated with Amivantamab IV): Switch from Amivantamab IV to SC-CF (Q2W); Cohort 5(Exon19del/Exon21 L858R NSCLC, 1L, Previously Untreated): Amivantamab (Q4W) + Lazertinib; Cohort6(Exon19del/Exon21L858R,NSCLC1L,PreviouslyUntreated):Amivantamab(Q2W)+Lazertinib+Anticoagulant
Drug: Carboplatin — Carboplatin will be administrated by IV infusion.
  Arms: Cohort 2(Exon20 NSCLC,1L, Previously Untreated): Amivantamab (Q3W) + Chemotherapy; Cohort 3(Exon19del/Exon21 L858R NSCLC,2L,Post Osimertinib):Amivantamab(Q3W)+Lazertinib+Chemotherapy; Cohort 3b(Exon19del/Exon21 L858R NSCLC, 2L, Post Osimertinib): Amivantamab (Q3W)+Chemotherapy; Cohort 7(Exon19del/Exon21 L858R NSCLC,2L,Post Amivantamab+Lazertinib):Amivantamab(Q3W)+Chemotherapy
Drug: Pemetrexed — Pemetrexed will be administered by IV infusion.
  Arms: Cohort 2(Exon20 NSCLC,1L, Previously Untreated): Amivantamab (Q3W) + Chemotherapy; Cohort 3(Exon19del/Exon21 L858R NSCLC,2L,Post Osimertinib):Amivantamab(Q3W)+Lazertinib+Chemotherapy; Cohort 3b(Exon19del/Exon21 L858R NSCLC, 2L, Post Osimertinib): Amivantamab (Q3W)+Chemotherapy; Cohort 7(Exon19del/Exon21 L858R NSCLC,2L,Post Amivantamab+Lazertinib):Amivantamab(Q3W)+Chemotherapy
Drug: Direct Oral Anticoagulant (DOAC) — DOAC will be administered orally.
  Arms: Cohort6(Exon19del/Exon21L858R,NSCLC1L,PreviouslyUntreated):Amivantamab(Q2W)+Lazertinib+Anticoagulant
Drug: Low Molecular Weight Heparin (LMWH) — LMWH will be administered subcutaneously.
  Arms: Cohort6(Exon19del/Exon21L858R,NSCLC1L,PreviouslyUntreated):Amivantamab(Q2W)+Lazertinib+Anticoagulant

SUMMARY:
The purpose of this study is to assess the anti-tumor activity and safety of amivantamab which will be administered as a co-formulation with recombinant human hyaluronidase PH20 (rHuPH20) (subcutaneous co-formulation [SC-CF]) in combination treatment (all cohorts except Cohort 4) and to characterize the safety of amivantamab SC-CF (Cohort 4).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed, locally advanced or metastatic, non-small cell lung cancer (NSCLC) that is not amenable to curative therapy including surgical resection or chemoradiation. Additional Cohort specific disease requirements include: Cohorts 1, 3, 3b, 5, 6 and 7: epidermal growth factor receptor (EGFR) exon 19 deletion (Exon19del) or Exon 21 L858R mutation; Cohort 2: EGFR Exon 20ins mutation. Cohorts 1,5,and6: Participant should not have received any prior systemic therapy for locally advanced or metastatic NSCLC. Cohort 2: Participant should not have received any prior systemic therapy for locally advanced or metastatic NSCLC. Cohorts 3and3b: Participant must have progressed on or after osimertinib monotherapy as the most recent line of treatment. Osimertinib must have been administered as either the first-line treatment for locally advanced or metastatic disease or in the second-line setting after prior treatment with first- or second-generation EGFR tyrosine kinase inhibitor (TKI) as a monotherapy. Cohort 4: Participants need to currently be on an amivantamab IV Q2W regimen (1,050 mg or 1,400 mg depending on weight) for at least 8 weeks, as part of standard of care, an expanded access program, or as a rollover from a long-term extension, without any amivantamab dose reduction. Cohort 7: Participants must have progressed on or after the combination of amivantamab and lazertinib as the most recent line of treatment. The combination of amivantamab and lazertinib must have been administered as the first-line treatment for locally advanced or metastatic disease. Cohort 2, 3, 3b, and 7 only: Squamous NSCLC are excluded. EGFR mutation must have been identified as determined by Food and Drug Administration (FDA) approved or other validated test of either circulating tumor deoxyribonucleic acid (ctDNA) or tumor tissue in a clinical laboratory improvement amendments (CLIA) certified laboratory (sites in the United states [US]) or an accredited local laboratory (sites outside of the US). A copy of the initial test report documenting the EGFR mutation must be included in the participant records and a deidentified copy must also be submitted to the sponsor
* All cohorts except Cohort 4: Participants must have at least 1 measurable lesion, according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. If the only target lesion has been previously irradiated, it must show signs of disease progression since radiation was completed If only 1 non-irradiated measurable lesion exists, which undergoes a biopsy and is acceptable as a target lesion, the baseline tumor assessment scans should be performed at least 14 days after the biopsy
* May have a prior or concurrent second malignancy (other than the disease under study) which natural history or treatment is unlikely to interfere with any study endpoints of safety or the efficacy of the study treatment(s)
* Have adequate organ (renal, hepatic, hematological, coagulation and cardiac) functions
* Participant must have eastern cooperative oncology group (ECOG) status of 0 or 1
* Cohort 6: Must be eligible for, and agree to comply with, the use of prophylactic anticoagulation with a direct oral anticoagulant or a low molecular weight heparin during the first 4 months of study treatment
* A participant must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of 6 months after receiving the last dose of study treatment. Participants with child bearing potential should consider preservation of eggs prior to study treatment as anti-cancer treatments may impair fertility

Exclusion Criteria:

* Participant has a medical history of interstitial lung disease (ILD), including drug induced ILD or radiation pneumonitis
* Participant has a history of hypersensitivity to any excipients of the investigational products to be used in their enrollment cohort
* Participant has received a live or live attenuated vaccine within 3 months before Cycle 1 Day 1. The seasonal influenza vaccine and non-live vaccines against Coronavirus disease 19 (COVID-19) are not exclusionary
* For all cohorts (with regimens potentially including lazertinib): Participant is currently receiving medications or herbal supplements known to be potent Cytochrome (CYP3A4/5) inducers and is unable to stop use for an appropriate washout period prior to Cycle 1 Day 1
* Other clinically active liver disease of infectious origin
* Participant has a history of clinically significant cardiovascular disease including, but not limited to: a) All cohorts: diagnosis of deep vein thrombosis or pulmonary embolism within 1 month prior to the first dose of study treatment(s), or any of the following within 6 months prior to the first dose of study treatment(s): myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary/peripheral artery bypass graft, or any acute coronary syndrome. Clinically non-significant thrombosis, such as non-obstructive catheter-associated clots, are not exclusionary; b) All cohorts (with regimens potentially including lazertinib): Participant has a significant genetic predisposition to venous thromboembolic events (VTE; such as Factor V Leiden); c) All cohorts (with regimens potentially including lazertinib): Participant has a prior history of VTE and is not on appropriate therapeutic anticoagulation as per NCCN or local guidelines; d) prolonged corrected QT interval by Fridericia (QTcF) interval greater than (>) 480 milliseconds (msec) or clinically significant cardiac arrhythmia or electrophysiologic disease (example, placement of implantable cardioverter defibrillator or atrial fibrillation with uncontrolled rate); e) uncontrolled (persistent) hypertension: systolic blood pressure >160 millimeter(s) of mercury (mmHg); diastolic blood pressure >100 mmHg; f) Congestive heart failure defined as NYHA class III-IV or hospitalization for congestive heart failure (CHF) (any New York Heart Association [NYHA] class) within 6 months of treatment initiation at Cycle 1/day 1 (C1D1); g) pericarditis/clinically significant pericardial effusion; h) myocarditis; i) baseline left ventricular ejection fraction (LVEF) below the institution's lower limit of normal at screening, as assessed by echocardiogram or multigated acquisition (MUGA) scan
* Participant has symptomatic brain metastases. A participant with asymptomatic or previously treated and stable brain metastases may participate in this study. Participants who have received definitive radiation or surgical treatment for symptomatic or unstable brain metastases and have been clinically stable and asymptomatic for at least 2 weeks before Screening are eligible, provided they have been either off corticosteroid treatment or are receiving low-dose corticosteroid treatment (less than or equal to [<=] 10 milligrams per day [mg/day] prednisone or equivalent) for at least 2 weeks prior to treatment allocation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2027-08-17 (Estimated); Study Completion 2027-08-17 (Estimated)

PRIMARY OUTCOMES:
All Cohorts Except Cohort 4: Objective Response Rate (ORR) Based on Investigator Assessment (INV) | Up to 1 year 6 months
  ORR based on INV will be reported. ORR is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR), based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, as determined by investigator.
Cohort 4: Number of Participants with Adverse Events (AEs) | Up to approximately 4 years and 9 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Cohort 4: Number of Participants with AEs by Severity | Up to approximately 4 years and 9 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Cohort 4: Number of Participants with Abnormalities in Clinical Laboratory Values | Up to approximately 4 years and 9 months
  Number of participants with abnormalities in clinical laboratory values (which includes serum chemistry, hematology, coagulation, urinalysis, and serology) will be reported.
Cohort 4: Number of Participants with Abnormalities in Clinical Laboratory Values by Severity | Up to approximately 4 years and 9 months
  Number of participants with laboratory values abnormalities which includes serum chemistry, hematology, coagulation, urinalysis, and serology) by severity will be reported. Severity of laboratory values abnormalities will be graded according to the NCI-CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.

SECONDARY OUTCOMES:
All Cohorts Except Cohort 4: Number of Participants with AEs | Up to 1 year 6 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
All Cohorts Except Cohort 4: Number of Participants with AEs by Severity | Up to 1 year 6 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
All Cohorts Except Cohort 4: Number of Participants with Abnormalities in Clinical Laboratory Values | Up to 1 year 6 months
  Number of participants with abnormalities in clinical laboratory values (which includes serum chemistry, hematology, coagulation, urinalysis, and serology) will be reported.
All Cohorts Except Cohort 4: Number of Participants with Abnormalities in Clinical Laboratory Values by Severity | Up to 1 year 6 months
  Number of participants with abnormalities in clinical laboratory values which includes serum chemistry, hematology, coagulation, urinalysis, and serology) by severity will be reported. Severity of laboratory values abnormalities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
All Cohorts Except Cohort 4: ORR Based on Independent Central Review (ICR) | Up to 1 year 6 months
  ORR based on ICR will be reported. The ORR is defined as the percentage of participants who achieve a CR or PR, based on RECIST version 1.1, as confirmed by ICR.
All Cohorts Except Cohort 4: Duration of Response (DoR) Based on Investigator Assessment (INV) | Up to 1 year 6 months
  DoR based on INV is defined as the time from the date of first documented response (PR or CR) until the date of documented progression or death, whichever comes first, for participants who have PR or CR.
All Cohorts Except Cohort 4: Time to Response (TTR) Based on INV | Up to 1 year 6 months
  TTR (that is, time to first response) based on INV is defined as the time from the first dose of study treatment to the date of first documentation of a response (PR or CR) prior to any disease progression and subsequent anticancer therapy, based on RECIST version 1.1., for participants who have PR or CR as their best response.
All Cohorts Except Cohort 4: Clinical Benefit Rate (CBR) | Up to 1 year 6 months
  CBR is defined as the percentage of participants achieving CR or PR, or durable standard deviation (SD) of a duration of at least 11 weeks as defined by RECIST version 1.1.
All Cohorts Except Cohort 4: Progression-free Survival (PFS) | Up to 3 years
  The PFS is defined as the time from the first dose of study treatment until the date of objective disease progression or death, whichever comes first, based on RECIST version 1.1.
All Cohorts Except Cohort 4: Overall Survival (OS) | Up to approximately 4 years
  The OS is defined as the time from the first dose of study treatment until the date of death due to any cause.
All Cohorts Except Cohort 4: Number of Participants with Venous Thromboembolic Events (VTE) | Up to 1 year 6 months
  Number of participants with adverse events of VTE (pulmonary embolism and deep vein thrombosis) will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
All Cohorts Except Cohort 4: Number of Participants with Venous Thromboembolic Events (VTE) by Severity | Up to 1 year 6 months
  Number of participants with adverse events of VTE (pulmonary embolism and deep vein thrombosis) by severity will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death).
All Cohorts Except Cohort 4: Serum Concentration Immediately Prior to the Next Dose Administration (Ctrough) of Amivantamab | Cycle 2 Day 1 of 28-day cycle
  Ctrough is defined as the serum concentration of amivantamab immediately prior to the next drug administration.
Cohort 4: Cancer Therapy Satisfaction as Assessed by Modified Therapy Administration Satisfaction Questionnaire - Intravenous (TASQ-IV) | Up to 1 year 6 months
  Patient-reported outcome (PRO): Cancer therapy satisfaction will be assessed using the modified TASQ-IV. The modified TASQ is a 12-item questionnaire measuring the impact of each mode of treatment administration on five domains: physical impact, psychological impact, impact on activities of daily living, convenience, and satisfaction. Each of the domain/scale scores is scored on a 1-100 scale, where 0 is worst and 100 is best.
Cohort 4: Cancer Therapy Satisfaction as Assessed by Modified Therapy Administration Satisfaction Questionnaire - Subcutaneous (TASQ-SC) | Up to 1 year 6 months
  PRO: Cancer therapy satisfaction will be assessed using the modified TASQ-SC. The modified TASQ is a 12-item questionnaire measuring the impact of each mode of treatment administration on five domains: physical impact, psychological impact, impact on activities of daily living, convenience, and satisfaction. Each of the domain/scale scores is scored on a 1-100 scale, where 0 is worst and 100 is best.
Cohort 4: Patient-reported Status as Assessed by Patient Global Impression of Change (PGIC) Scale Score | Up to 1 year 6 months
  Patient-reported status as assessed by PGIC scale score will be reported. The PGIC is an assessment of the participant's overall sense of whether there has been a change since starting treatment. The PGIC is a 7-point response scale. Participants will be asked to rate their current fatigue as compared to when they started the study, using the following 7-point scale: 1 = Much better, 2 = Moderately better, 3 = A little better, 4 = No change, 5 = A little worse, 6 = Moderately worse, and 7 = Much worse.
Cohort 4: Patient-reported Status as Assessed by Patient Global Impression of Symptom Severity (PGIS) Scale Score | Up to 1 year 6 months
  Patient-reported status as assessed by PGIS scale score will be reported. The PGIS is an assessment of lung cancer severity at a given point in time. The PGIS is a 5-point response scale. Participants will be asked to rate their fatigue over the past 7 days using the following 5-point scale: 1 = None, 2 = Mild, 3 = Moderate, 4 = Severe, and 5 = Very severe.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (109):
- United States (25):
  - University of California at San Diego, La Jolla, California
  - University of California Irvine, Orange, California
  - Stanford Cancer Institute, Stanford, California
  - Johns Hopkins Office of Capital Region Research - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Baptist Lynn Cancer Institute, Boca Raton, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth, Orlando, Florida
  - H. Lee Moffitt Cancer & Research Institute, Tampa, Florida
  - University of Kansas Cancer Center, Westwood, Kansas
  - Sidney Kimmel Cancer Center - Bayview Campus, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Washington University School Of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Hematology-Oncology Associates of CNY, East Syracuse, New York
  - Novant Health, Charlotte, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Cleveland Clinic, Mayfield Heights, Ohio
  - Cleveland Clinic, Warrensville Heights, Ohio
  - The Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
- Brazil (9):
  - Fundacao Pio XII, Barretos
  - PERSONAL Oncologia de Precisao e Personalizada, Belo Horizonte
  - Instituto do Cancer de Londrina Hospital do Cancer de Londrina, Londrina
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Instituto D Or de Pesquisa e Ensino IDOR, Rio de Janeiro
  - Instituto D Or de Pesquisa e Ensino IDOR, Salvador
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Impar Servicos Hospitalares SA Hospital Nove de Julho, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
- China (18):
  - Affiliated Hospital of Hebei University, Baoding
  - Jilin cancer hospital, Changchun
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - The First Affiliated Hospital of PLA Army Medical University, Chongqing
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Huizhou Municipal Central Hospital, Huizhou
  - Liuzhou people's Hospital, Liuchow
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Hospital of Jiangnan University, Wuxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
- France (6):
  - Centre Francois Baclesse, Caen
  - Centre Georges-François Leclerc, Dijon
  - Institut de Cancérologie du Gard, Nîmes
  - Institut Curie, Paris
  - Institut de cancerologie de l'ouest, Saint-Herblain
  - Gustave Roussy, Villejuif
- Germany (5):
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitaetsklinikum Koelnt, Cologne
  - LungenClinic Grosshansdorf GmbH, Grosshandorf
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikum Würzburg Mitte gGmbH Standort Missioklinik, Würzburg
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (5):
  - Policlinico Hospital San Martino- IRCCS for Oncology, Genova
  - Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Azienda Ospedaliera Specialistica dei Colli, Naples
- Japan (6):
  - National Hospital Organization Himeji Medical Center, Himeji
  - Matsusaka Municipal Hospital, Matsusaka
  - Niigata Cancer Center Hospital, Niigata
  - Shizuoka Cancer Center, Shizuoka
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Malaysia (4):
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak, Kuching
  - Beacon Hospital Sdn Bhd, Petaling Jaya
- South Korea (5):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (14):
  - Hosp Univ A Coruna, A Coruña
  - General University Hospital of Alicantet, Alicante
  - Hosp. Del Mar, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Virgen Macarena, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Gral. Univ. Valencia, Valencia
- United Kingdom (7):
  - Cheltenham General Hospital, Cheltenham
  - Torbay Hospital-Devon, Devon
  - Edinburgh Cancer Centre Western General, Edinburgh
  - Leicester Royal Infirmary, Leicester
  - University College London Hospitals, London
  - Nottingham City Hospital, Nottingham
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency